CLINICAL TRIAL: NCT02719704
Title: Effect of a Multicomponent Intervention Program on Physical Fitness Related to Health and Body Image: School-based Study With Adolescents of Florianópolis, Santa Catarina, Brazil
Brief Title: School-based Multicomponent Intervention on Physical Fitness Related to Health and Body Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Catarina Federal University (Other)
Responsible Party: Principal Investigator, Giseli Minatto, PhD Student, Universidade Federal de Santa Catarina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEXA-SE
Record Dates: First submitted 2016-02-29; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Physical Fitness; Body Image

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "MEXA-SE" (Experimental): Intervention on physical fitness, eating habits and body image
  Interventions: Behavioral: "MEXA-SE"
- Control (No Intervention): School of the control group carried out one semester with the regular and traditional activities. The control school had three physical educations lessons per week, similar of experimental schools.
- "Espelho, espelho meu" (Experimental): School-based intervention on body image
  Interventions: Behavioral: "Espelho, espelho meu"

INTERVENTIONS:
Behavioral: "MEXA-SE" — MEXA-SE (move yourself) was structured into three main components: A) Physical fitness: The first component was to increase time in moderate to vigorous physical activity during Physical Education lessons. There were also prompts to help students to engage in increased physical activity during school recess; B) Eating habits: The second component consisted of six sessions (45 minutes per session) designed to promote reflection and positive changes in eating habits and health care (to improve knowledge and eating habits), conducted by nutritionist; C) Body image: The third component was composed of 3 sessions (45 minutes per session) focused on body image satisfaction ("Espelho, espelho meu": School based Intervention) conducted by Physical Education researcher.
  Arms: "MEXA-SE"
Behavioral: "Espelho, espelho meu" — Behavioral: "Espelho, espelho meu": School based intervention on body image. Body image is worked in four 45 minutes sessions, conducted with a frequency of once a week by a researcher. The topics covered in these sessions refer to: Beauty Standards (media influence and formation of body image), individual qualities (individual and classmates qualities) and selfesteem. These meetings will be held through video, lecture, dynamics, photo sessions and preparation of posters.
  Arms: "Espelho, espelho meu"

SUMMARY:
The main purpose of this study is to analyse the effect of a multicomponent intervention, applied during one scholar semester, on body composition, strength, flexibility, cardiorespiratory fitness, lipid and metabolic profile, and body image of students from sixth to ninth grade. This is a non-randomized controlled design. Approximately 568 schoolchildren of grades sixth through ninth were recruited from 2 public secondary schools in Florianópolis, Brazil. The main component of the intervention entitled "MEXA-SE" (move yourself) consisted of the implementation of three physical education classes per week with aerobic exercises, strength and flexibility activities. In addition, play activities in school recess, and educational activities on physical activity, sedentary behaviour, eating habits and body image were performed. Data collection was performed before and immediately after 14 weeks of intervention. The primary outcomes included the body composition, strength, flexibility, cardiorespiratory fitness, lipid and metabolic profile, and body image. Other variables included were: physical activity level, sedentary behaviour, and blood pressure level. Other components of the lifestyle (e.g., eating habits), psychological (e.g., self-rated health) also were evaluated in the participants. Descriptive analysis, two-way ANOVA for mixed models and ANCOVA will be applied for within and between comparison groups, if the premises of this test are met. The level of significance for the study was 5% for two-tailed tests.

ELIGIBILITY:
Inclusion Criteria:

* Students volunteering as participation;
* Students regularly enrolled from the 6th to the 9th grades in the Florianópolis municipal school system.

Exclusion Criteria:

* Students of other grades;
* Students who dropout of school;
* Students with incomplete data at baseline and end 14 weeks;
* Students who are absence in the school days of data collection;
* Students who refused to participate in data collection or intervention;

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 568 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change on body mass index | Baseline, 14 weeks
  Anthropometric measurements of body mass (kilograms), height (centimeters) to calculate body mass index (kilograms per square meter).
Change on skinfold thickness | Baseline, 14 weeks
  Anthropometric measurements of skinfold thickness (millimeters) of biceps, triceps, subscapular, iliac crest and medial calf.
Change on flexibility | Baseline, 14 weeks
  Modified Sit and Reach test (centimeters).
Change on muscular strength | Baseline, 14 weeks
  Handgrip test measured by dynamometer (Kilograms).
Change on resistance levels | Baseline, 14 weeks
  Modified abdominal test (number of repetitions).
Change on cardiorespiratory fitness | Baseline, 14 weeks
  20-m shuttle run test (laps).
Change on body image | Baseline, 14 weeks
  Self-perception (questionnaire).
Change on lipid | Baseline, 14 weeks
  Enzymatic colorimetric test
Change on girth | Baseline, 14 weeks
  Anthropometric measurements of girth (centimeters) of relaxed arm and waist.
Change on glucose profile | Baseline, 14 weeks
  Enzymatic colorimetric test
Change on percent body fat | Baseline, 14 weeks
  Measurement by bioelectrical impedance.
Change on fat free mass | Baseline, 14 weeks
  Measurement by bioelectrical impedance.
Change on percent of water | Baseline, 14 weeks
  Measurement by bioelectrical impedance.
Change on resistance | Baseline, 14 weeks
  Measurement by bioelectrical impedance.
Change on reactance | Baseline, 14 weeks
  Measurement by bioelectrical impedance.

SECONDARY OUTCOMES:
Change on physical activity at school | Baseline, 14 weeks
  ActiGraph accelerometers.
Change on leisure physical activity | Baseline, 14 weeks
  List of physical activities practiced last week indicating the frequency and duration, commuting to school and preferred leisure activities reported in guided questionnaire.
Change on sedentary behaviour (television time) | Baseline, 14 weeks
  Time in front of television during the week and over the weekend reported in guided questionnaire.
Change on sedentary behaviour (computer time) | Baseline, 14 weeks
  Time in computer and / or video games during the week and over the weekend reported in guided questionnaire.
Change on blood pressure levels | Baseline, 14 weeks
  Measured by Automatic blood pressure monitor.
Food consumption | Baseline, 14 weeks
  Food consumption reported in guided questionnaire.
Food Knowledge | Baseline, 14 weeks
  Knowledge consumption reported in guided questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Edio Luiz Petroski, Doctor, Study Director — Federal University of Santa Catarina; Cilene Rebolho Martins, PhD Student, Principal Investigator — Federal University of Santa Catarina; Juliane Berria, PhD Student, Principal Investigator — Federal University of Santa Catarina; Giseli Minatto, PhD Student, Principal Investigator — Federal University of Santa Catarina; Luiz R. A. de Lima, PhD Student, Principal Investigator — Federal University of Santa Catarina; Jéssika A. J. Vieira, Master Degree Student, Principal Investigator — Federal University of Santa Catarina; André Machado, Master Degree Student, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- Federal University of Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Martins PC, de Lima LRA, Berria J, Petroski EL, da Silva AM, Silva DAS. Association between phase angle and isolated and grouped physical fitness indicators in adolescents. Physiol Behav. 2020 Apr 1;217:112825. doi: 10.1016/j.physbeh.2020.112825. Epub 2020 Jan 25. PMID 31991158